CLINICAL TRIAL: NCT00311441
Title: A Phase IV, Randomized, Controlled, Single-Blind, Multi-Center Study in Children to Evaluate the Safety, Tolerability and Immunogenicity of Two TBE Vaccines Administered According to Two Different Schedules.
Brief Title: Study of the Safety, Tolerability and Immune Response of TBE Vaccines Administered to Healthy Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Collaborators: Novartis Vaccines (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: M48P3; 911
Record Dates: First submitted 2006-04-03; First posted 2006-04-06 (Estimated); Last update posted 2008-03-17 (Estimated); Status verified 2008-03

CONDITIONS: Encephalitis, Tick-Borne
Keywords: TBE, children, vaccine
MeSH Terms: conditions — Encephalitis, Tick-Borne

INTERVENTIONS:
Biological: Tick-Borne Encephalitis vaccine

SUMMARY:
The purpose of this study is to evaluate the safety, immunogenicity and tolerability of TBE vaccines administered to children.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female children, 1 to 10 years of age.

Exclusion Criteria:

* Subjects with documented evidence of TBE
* Subjects, who have been previously vaccinated against TBE

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 300
Dates: Start 2005-03

PRIMARY OUTCOMES:
Immunogenicity of two pediatric TBE vaccines as measured by neutralization test and ELISA on days 28, 42, 300, and 321.

SECONDARY OUTCOMES:
Tolerability of two paediatric TBE vaccines with respect to local and systemic reactions including fever

CONTACTS AND LOCATIONS:
Overall Officials: Drug Information Services, Study Director — Novartis Vaccines & Diagnostics
Locations (1):
- Weilheim, Germany